CLINICAL TRIAL: NCT01839851
Title: Evaluation of Hair Cortisol in Patients With Asthma or Allergic Rhinitis Treated With Topical (Inhaled or Intranasal) Corticosteroids
Brief Title: Hair Cortisol in Asthma or Allergic Rhinitis Treated With Topical Corticosteroids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC-13-0047-CTIL
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2013-10

CONDITIONS: ASTHMA; ALLERGIC RHINITIS
Keywords: Hair cortisol; asthma; allergic rhinitis; inhaled corticosteroids; intranasal glucocorticoids
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — Therapeutics; Budesonide, Formoterol Fumarate Drug Combination; Beclomethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asthma: Treatment with any inhaled corticosteroid
  Interventions: Drug: Treatment with any inhaled corticosteroid
- Allergic rhinitis: Treatment with any intranasal glucocorticoid
  Interventions: Drug: Treatment with any intranasal glucocorticoid
- Asthma and allergic rhinitis: Inhaled corticosteroid + intranasal glucocorticoid
  Interventions: Drug: Treatment with any inhaled corticosteroid; Drug: Treatment with any intranasal glucocorticoid

INTERVENTIONS:
Drug: Treatment with any inhaled corticosteroid — Use of any inhaled corticosteroid (daily frequency and dose will be registered)
  Other Names: Symbicort; Budicort; Qvar
  Groups: Asthma; Asthma and allergic rhinitis
Drug: Treatment with any intranasal glucocorticoid — Use of any inhaled intranasal glucocorticoid (daily dose and frequency will be registered)
  Other Names: Steronase
  Groups: Allergic rhinitis; Asthma and allergic rhinitis

SUMMARY:
The purpose of this study is to prospectively examine the relation between topical corticosteroid use and hair cortisol concentration, among patients with moderate persistent asthma or allergic rhinitis. The investigators hypothesize that patients with asthma or allergic rhinitis treated with topical corticosteroids (i.e. inhaled corticosteroids (ICS) or intranasal glucocorticoids (INGC)) have higher levels of hair cortisol after 3 months of treatment than during the 3 months prior to initiation of treatment.

DETAILED DESCRIPTION:
Inhaled corticosteroids have proven effective in the treatment of asthma, suppressing airway inflammation and reducing bronchial hyper-responsiveness. Beneficial clinical outcomes include fewer asthmatic symptoms, increased lung function, improved asthma-specific quality of life, and fewer asthmatic exacerbations, including severe attacks resulting in hospitalization or death. ICS are commonly used when asthmatic episodes are too frequent or too severe to be controlled solely by short acting beta agonists. ICS have few adverse effects at low to medium doses, which are mainly local effects such as hoarseness and oral thrush. On the other hand, high doses of ICS are associated with systemic effects such as increased risk of skin bruising, cataracts, elevated intraocular pressure and accelerated loss of bone mass. While there is less evidence pointing towards systemic effects of low to medium doses of ICS, several studies have suggested that such an effect exists. One study demonstrated changes in the hypothalamic-pituitary-adrenal (HPA) axis with ICS administration at doses as low as 88 μg of fluticasone per day. Moreover, a study in children showed ICS did not influence basal cortisol levels but significantly reduced peak cortisol and adrenocorticotropic hormone levels.

Hence, the extent of the systemic effect of ICS at high doses and especially at low to medium doses is not fully understood. This is partly due to the nature of most of the systemic side-effects which necessitate long term follow-up of a large population of patients, but also because of technical difficulties in assessing systemic cortisol levels over a prolonged period of time.

A similar clinical conundrum exists with intranasal glucocorticoids (INGC), regarding their systemic effect. INGCs are considered the first-line of medical therapy for allergic rhinitis and are more effective than systemic antihistamines. The most common adverse effects stem from local irritation of the nasal mucosa, while systemic effects are much rarer. The effect of INGC on the HPA axis and growth has been evaluated extensively in children. Most studies, especially those with the second generation agents and recommended doses, showed no or limited HPA suppression. Despite these reassuring data, the adverse effects of INGC can be additive with those of other glucocorticoid preparations for comorbid conditions, and thus caution should be exercised. A handful of studies have demonstrated detrimental effects of INGC therapy on bone mineral density and intraocular pressure. These studies have small sample sizes and have not clearly proven whether these effects result in clinically relevant long term outcomes, such as fractures. As a result, these studies are not reflected in current practice guidelines.

Cortisol levels are routinely determined from blood, salivary or urinary samples However, these methods do not provide information on long term cortisol secretion, accounting for the variability of HPA axis activity. There is a growing pool of evidence that shows that Hair Cortisol Concentration (HCC) examination provides a reliable retrospective estimation of integrated cortisol secretion over a period of several months. Hair grows at a rate of about 1 cm/month, thus 3 cm of hair would give an indication of the cortisol levels over the previous 3 months. HCC correlates with 24h urinary cortisol levels, but not with salivary or serum cortisol, supporting use of HCC as an indicator of cortisol levels over time rather than a point measurement. HCC has been evaluated in several clinical settings in which activity of the HPA axis and cortisol levels over a period of time are of interest. Studies have demonstrated increased levels of hair cortisol in patients with stress as well as in conditions associated with stress such as pregnancy, unemployment, PTSD, alcohol withdrawal, chronic pain and myocardial infarction. Elevated levels of hair cortisol were also shown in Cushing's syndrome, with reduced levels after correction of the disorder.

No study to date has examined the correlation between the use of inhaled or intranasal corticosteroids and levels of cortisol in hair. If such a correlation exists, it would indicate systemic absorption of these topical steroids which in turn would suggest a potential for systemic side effects. In addition, and pending further studies, HCC may serve as a validated test to determine which patients are more prone to systemic side effects, as well as help in assessing compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Diagnosis of asthma or allergic rhinitis, or both.
* Planned initiation of treatment with ICS and/or INGC at study recruitment, according to routine clinical practice

Exclusion Criteria:

* Use of inhaled, systemic or topical corticosteroids at study initiation, or during the previous 6 months.
* Use of topical corticosteroid ointments or cream, or systemic corticosteroids during the study period.
* Disorders associated with disruption of HPA axis (Cushing syndrome, Addison syndrome).
* Insufficient hair for analysis
* Bleaching or use of artificial hair color.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with asthma or allergic rhinitis requiring treatment with topical corticosteroids (inhaled corticosteroids or intranasal glucocorticoids), presenting to the Meir Medical Center Allergy and Immunology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in concentration of hair cortisol under topical corticosteroid treatment | Hair cortisol concentration 3 months after initiation of treatment with inhaled or intranasal corticosteroids compared to concentration of hair cortisol at study initiation
  The primary outcome will be evaluated separately in each of the three distinct study cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Eilon Krashin, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Stalder T, Kirschbaum C. Analysis of cortisol in hair--state of the art and future directions. Brain Behav Immun. 2012 Oct;26(7):1019-29. doi: 10.1016/j.bbi.2012.02.002. Epub 2012 Feb 15. PMID 22366690